CLINICAL TRIAL: NCT04446975
Title: Best Practice Alert for Post-Surgical Opioid Prescribing At Discharge
Brief Title: Best Practice Alert for Opioid Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Nebraska (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 19-3095
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use

STUDY DESIGN:
Intervention Model Description: This trial will be designed using a stepped wedge design with randomization occurring based on timing and location of enrollment according to PRECIS-2 (PRagmatic Explanatory Continuum Indicator Summary) to maximize applicability. The BPA will be turned "OFF" vs. "ON" in the participating hospitals according to each 8-week study interval. OFF and ON periods will be separated by 4-week washout intervals. An 8-week period prior to study start will provide baseline trends in prescription patterns. The investigation will commence with two "OFF" periods to assess if reduction in prescribing patterns occurs over time regardless of the intervention. Two "ON" periods at the end of the study will determine if any observed changes in prescribing patterns stabilize or continued changes take place.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPA Off (No Intervention): No best-practice alert (BPA) message is displayed to providers.
- BPA On (Experimental): BPA message is displayed to providers based on patient opioid intake as reported in the electronic health record (EHR).
  Interventions: Other: BPA

INTERVENTIONS:
Other: BPA — At the time of writing the prescription an automatic notification will appear on the care provider's screen that identifies a suggested post-discharge opioid dose within the electronic prescription pad. If approved by the provider, opioid-only prescriptions will be written as suggested. Final dosing decisions and drug choices will remain at the discretion of the treating provider.
  Arms: BPA On

SUMMARY:
The investigators will embed a developed decision support tool into the electronic health record (EHR) to individualize pain therapy in surgical patients after hospital discharge and test its performance in a pragmatic clinical trial.

Preliminary data indicate that current opioid prescription practice after surgery follows a "one size fits all" pattern. In-hospital opioid use prior to discharge serves as a reliable indicator to estimate needs for analgesic medications at home. The investigators will test the hypothesis that the existing tool will enable providers to write need-based prescriptions based on prior-to-discharge opioid use, empower patients to maximize alternatives to opioids (ALTO) therapies at home, while minimizing the need for rescue prescriptions. The investigators will test this tool prospectively in a cohort of ~1,000 providers (primary subjects) and ~39,000 surgical patients (secondary subjects) in four University of Colorado Health (UCHealth) hospitals (clusters to be exposed versus (vs.) non-exposed to the intervention).

DETAILED DESCRIPTION:
Converting knowledge on actual need for opioid pain medications after surgery into tangible benefits can prevent over-prescription of opioids that become available for non-medical use. The objective of this aim is to prescribe pain medications after surgery in a patient-centered fashion. The investigators have used the average amount of opioid medications (in milligram morphine equivalents - MME) taken prior to discharge to inform the clinical decision support tool. This tool will reduce the amount of opioid medications prescribed while maintaining patient post-operative pain control. The calculated "prior to discharge daily MME dose" will be applied to generate a recommendation for the prescription of a cumulative opioid dose that will be displayed when the electronic order entry for the post-discharge pain medication is made in the EHR using a best-practice alert (BPA). In addition, the provider will be prompted to also prescribe non-opioid analgesic medications. This BPA was developed by the Principal Investigator under guidance of the UCHealth System Multidisciplinary Opioid/Pain Management Committee as well as published guidelines.

Based on the relationship between opioids taken prior to discharge and post-discharge opioid intake described above as well as published guidelines for post-discharge prescriptions after surgery will use a tiered approach towards determining the total amount of opioids to be prescribed. Accordingly, the investigators have integrated an algorithm into the BPA such that opioid intake from the EHR only triggers the BPA if the total amount of prescribed opioids exceeds the predicted thresholds.

The opioid prescribing BPA will be assessed over a 44-week period in all eligible patients. At the time of writing the prescription an automatic notification will appear on the care provider's screen that identifies a suggested post-discharge opioid dose within the electronic prescription pad. If approved by the provider, opioid-only prescriptions will be written as suggested. Final dosing decisions and drug choices will remain at the discretion of the treating provider and will be tracked. The investigators will use an all "On" vs. all "Off" configuration to answer the questions if the average amount of total opioids per post-discharge prescription is lower with the BPA active. The investigation will commence with two "Off" periods to assess if reduction in prescribing patterns occurs over time regardless of the intervention. Two "On" periods at the end of the study will determine if any observed changes in prescribing patterns stabilize or continued changes take place.

ELIGIBILITY:
Inclusion Criteria:

Primary subjects:

• Credentialed providers (attending, fellow, and resident physicians, advanced practice providers including nurse practitioners and physician assistants) at each UCH (UC Health) site writing a discharge opioid prescription are eligible to receive the intervention.

Secondary subjects:

• Adult surgical inpatients age 18 and older within the UCHealth system at 4 different hospitals including UCH Metro, UCH Memorial Central, Medical Center of the Rockies, and Poudre Valley Hospital.

Exclusion Criteria:

Primary subjects:

• None

Secondary subjects:

• Less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21689 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Bartels, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Bartels K, Fernandez-Bustamante A, McWilliams SK, Hopfer CJ, Mikulich-Gilbertson SK. Long-term opioid use after inpatient surgery - A retrospective cohort study. Drug Alcohol Depend. 2018 Jun 1;187:61-65. doi: 10.1016/j.drugalcdep.2018.02.013. Epub 2018 Mar 27. PMID 29627407
- [Background] Chen EY, Marcantonio A, Tornetta P 3rd. Correlation Between 24-Hour Predischarge Opioid Use and Amount of Opioids Prescribed at Hospital Discharge. JAMA Surg. 2018 Feb 21;153(2):e174859. doi: 10.1001/jamasurg.2017.4859. Epub 2018 Feb 21. PMID 29238810

RESULTS

PARTICIPANT FLOW:
Groups:
- Site 1, BPA Off First; Site 4, BPA Off First: Treatment sequence:
  * BPA Off
  * Washout period
  * BPA On
  * Washout period
  * BPA Off
  * Washout period
  * BPA On
- Site 2, BPA On First; Site 3, BPA On First: Treatment sequence:
  * BPA On
  * Washout period
  * BPA Off
  * Washout period
  * BPA On
  * Washout period
  * BPA Off
Period: Randomization Period 1 (8 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 2435 | 1295 | 883 | 833
Completed | 2435 | 1295 | 883 | 833
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (4 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Randomization Period 2 (8 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 2527 | 1285 | 927 | 936
Completed | 2527 | 1285 | 927 | 936
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (4 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Randomization Period 3 (8 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 2174 | 1105 | 818 | 821
Completed | 2174 | 1105 | 818 | 821
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (4 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Randomization Period 4 (8 Weeks)
Arm/Group | Site 1, BPA Off First | Site 2, BPA On First | Site 3, BPA On First | Site 4, BPA Off First
Started | 2607 | 1248 | 963 | 832
Completed | 2607 | 1248 | 963 | 832
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BPA Off: No BPA message is displayed to providers.
- BPA On: BPA message is displayed to providers based on patient opioid intake as reported in the EHR.
  BPA: At the time of writing the prescription an automatic notification will appear on the care provider's screen that identifies a suggested post-discharge opioid dose within the electronic prescription pad. If approved by the provider, opioid-only prescriptions will be written as suggested. Final dosing decisions and drug choices will remain at the discretion of the treating provider.
- Total: Total of all reporting groups
Arm/Group | BPA Off | BPA On | Total
Number analyzed (Participants) | 10686 | 11003 | 21689
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (18.2) | 56.3 (18.1) | 56.5 (18.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4907 | 5137 | 10044
  Non Male | 5779 | 5866 | 11645
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 1468 | 1524 | 2992
  Ethnicity: Non-Hispanic | 9112 | 9368 | 18480
  Ethnicity: Unknown | 106 | 111 | 217
Region of Enrollment [Number; unit: participants]
  United States | 10686 | 11003 | 21689

OUTCOME MEASURES:

1. Primary Outcome: Opioids Prescribed at Discharge
Description: Prescribed milligram morphine equivalents (MME) discharge opioid dose as recorded in the electronic health record
Time Frame: 1 day, on discharge date from hospital
Measure: Median (Inter-Quartile Range); unit: miligram morphine equivalents
Arm/Group | BPA Off | BPA On
Number analyzed (Participants) | 10686 | 11003
miligram morphine equivalents | 100 [0 to 225] | 75 [0 to 225]

2. Secondary Outcome: Number of Participants With Opioid/Non-opioid Combination Medications Prescribed on Day of Discharge
Description: Number of Participants prescribed discharge non-opioid analgesic medications (opioid/non-opioid combination formulations) as recorded in the electronic health record
Time Frame: 1 day, on discharge date from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | BPA Off | BPA On
Number analyzed (Participants) | 10686 | 11003
Participants | 1758 | 1687

3. Secondary Outcome: Number of Participants With Opioid Prescriptions After Discharge
Description: Number of participants with opioid prescriptions after discharge as recorded in the electronic health record
Time Frame: "Day of discharge +1" until 28 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | BPA Off | BPA On
Number analyzed (Participants) | 10686 | 11003
Participants | 1870 | 2046

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Other Adverse Events were not monitored/assessed through study completion, an average of 28 days.
Description: All-Cause Mortality and Other Adverse Events were not monitored/assessed through study completion, an average of 28 days.
Arm/Group | BPA Off | BPA On
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT04446975/Prot_SAP_000.pdf